CLINICAL TRIAL: NCT01750281
Title: A Phase II, Double-Blind, Randomised, Placebo-Controlled Study to Assess the Efficacy and Safety of Selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate) in Combination With Docetaxel, Compared With Placebo in Combination With Docetaxel, in Patients Receiving Second Line Treatment for Locally Advanced or Metastatic Non Small Cell Lung Cancer (Stage IIIB - IV)
Brief Title: Assess Efficacy and Safety of AZD6244 in Combination With Docetaxel in Patients Receiving Second Line Non Small Cell Lung Cancer Treatment.
Acronym: SELECT-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1532C00064; 2012-003622-25 (EudraCT Number)
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Locally Advanced or Metastatic Non Small Cell Lung Cancer Stage IIIb - IV
Keywords: Mitogen-Activated Protein Kinase Kinase inhibitor; Non Small Cell Lung Cancer; Metastatic; Second line treatment for Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — AZD 6244; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Selumetinib 75 mg twice daily +Docetaxel 75 mg/m2 (Experimental): Selumetinib capsules will be administered orally uninterrupted twice daily in combination with docetaxel 75 mg/m2 intravenously administered on day 1 of each 21 day cycle.
  Interventions: Drug: Selumetinib 75 mg; Drug: Docetaxel 75 mg/m2
- Selumetinib 75 mg twice daily + Docetaxel 60 mg/m2 (Experimental): Selumetinib capsules will be administered orally uninterrupted twice daily in combination with docetaxel 60 mg/m2 intravenously administered on day 1 of each 21 day cycle.
  Interventions: Drug: Selumetinib 75 mg; Drug: Docetaxel 60 mg/m2
- Placebo twice daily + Docetaxel 75 mg/m2 (Experimental): Three placebo capsules will be administered orally uninterrupted twice daily in combination with docetaxel 75 mg/m2 intravenously administered on day 1 of each 21 day cycle.
  Interventions: Drug: Docetaxel 75 mg/m2; Drug: Placebo

INTERVENTIONS:
Drug: Selumetinib 75 mg — Three selumetinib capsules (Hyd-Sulfate) 25 mg will be administered orally, twice daily, (75 mg dose bd) on an uninterrupted schedule.
  Arms: Selumetinib 75 mg twice daily + Docetaxel 60 mg/m2; Selumetinib 75 mg twice daily +Docetaxel 75 mg/m2
Drug: Docetaxel 75 mg/m2 — Docetaxel 75 mg/m2 will be administered intravenously on day 1 of each 21 day cycle.
  Arms: Placebo twice daily + Docetaxel 75 mg/m2; Selumetinib 75 mg twice daily +Docetaxel 75 mg/m2
Drug: Docetaxel 60 mg/m2 — Docetaxel 60 mg/m2 will be administered intravenously on day 1 of each 21 day cycle.
  Arms: Selumetinib 75 mg twice daily + Docetaxel 60 mg/m2
Drug: Placebo — Three placebo capsules will be administered orally uninterrupted twice daily.
  Arms: Placebo twice daily + Docetaxel 75 mg/m2

SUMMARY:
The purpose of this study is to treat patients with locally advanced or metastatic NSCLC with a combination therapy of selumetinib and two different doses of docetaxel 75mg/m2 or 60 mg/m2 vs placebo and compare how well each dose affects how their cancer responds. It will also help us to understand the tolerability profile of the different dosing regimens in these patients

DETAILED DESCRIPTION:
A Phase II, Double-Blind, Randomised, Placebo-Controlled Study to Assess the Efficacy and Safety of Selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate) in Combination with Docetaxel, Compared with Placebo in Combination with Docetaxel, in Patients receiving second line treatment for Locally Advanced or Metastatic Non Small Cell Lung Cancer (Stage IIIB - IV)

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures
* Male or female, aged 18 years or older
* Histological or cytological confirmation of locally advanced or metastatic NSCLC (IIIB-IV)
* Prospective confirmation of KRAS mutation negative status as determined via an AZ approved laboratory
* Failure of 1st line anti-cancer therapy due to radiological documentation of disease progression in advanced disease or subsequent relapse of disease following 1st line therapy

Exclusion Criteria:

* Mixed small cell and non-small cell lung cancer histology
* Received >1 prior anti-cancer drug regimen for advanced or metastatic NSCLC. Patients who develop disease progression while on switch maintenance therapy (maintenance using an agent not in the first-line regimen) will not be eligible.
* Other concomitant anti-cancer therapy agents except steroids
* Prior treatment with a MEK (Mitogen-Activated Protein Kinase) inhibitor or any docetaxel-containing regimen (prior treatment with paclitaxel is acceptable)
* The last radiation therapy within 4 weeks prior to starting study treatment, or limited field of radiation for palliation within 7 days of the first dose of study treatment.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2012-12-18 (Actual); Primary Completion 2016-01-27 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Mariani, MD, Study Chair — AstraZeneca UK, MSD; Pasi Janne, MD, Principal Investigator — Dana-Farber Cancer Institute, USA; Jean-Charles Soria, MD, Principal Investigator — Institut de Cancerology Gustave Roussy, France
Locations (56):
- United States (12):
  - Research Site, Santa Monica, California
  - Research Site, Aurora, Colorado
  - Research Site, Hollywood, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Marrero, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
- Brazil (7):
  - Research Site, Barretos
  - Research Site, Brasília
  - Research Site, Ijuí
  - Research Site, Porto Alegre
  - Research Site, Santo André
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (4):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Vratsa
- France (6):
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Clermont-Ferrand
  - Research Site, Lille
  - Research Site, Pierre-Bénite
  - Research Site, Villejuif
- Germany (8):
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Großhansdorf
  - Research Site, Karlsruhe
  - Research Site, Löwenstein
  - Research Site, Moers
  - Research Site, Wiesbaden
  - Research Site, Würzburg
- Hungary (8):
  - Research Site, Budapest
  - Research Site, Edelény
  - Research Site, Győr
  - Research Site, Kaposvár
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Székesfehérvár
  - Research Site, Törökbálint
- Netherlands (4):
  - Research Site, 's-Hertogenbosch
  - Research Site, Amsterdam
  - Research Site, Bergen op Zoom
  - Research Site, Maastricht
- Poland (7):
  - Research Site, Gdansk
  - Research Site, Grudziądz
  - Research Site, Krakow
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Sucha Beskidzka
  - Research Site, Szczecin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Soria JC, Fulop A, Maciel C, Fischer JR, Girotto G, Lago S, Smit E, Ostoros G, Eberhardt WEE, Lishkovska P, Lovick S, Mariani G, McKeown A, Kilgour E, Smith P, Bowen K, Kohlmann A, Carlile DJ, Janne PA. SELECT-2: a phase II, double-blind, randomized, placebo-controlled study to assess the efficacy of selumetinib plus docetaxel as a second-line treatment of patients with advanced or metastatic non-small-cell lung cancer. Ann Oncol. 2017 Dec 1;28(12):3028-3036. doi: 10.1093/annonc/mdx628. PMID 29045535
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1532C00064&attachmentIdentifier=fcbb09ba-0d2c-4d3b-8b1b-962bedef9990&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initially the study protocol allowed patients with KRASm (KRAS mutation positive), KRAS NMD (No mutation detected) and KRAS mutation status unknown. Recruitment was put on hold after the 77th patient was randomised in September 2013, to allow a protocol amendment to include only patients with centrally confirmed KRAS NMD NSCLC to be enrolled.
Pre-assignment Details: The Protocol Section "Enrolment Number" of 466 includes 1 patient who was pre-screened twice. Of the 465 unique "pre-screened" patients, 337 gave informed consent and of these, 212 were randomised. 211 received at least 1 dose of treatment and were included in the safety analysis set. Patients received selumetinib (AZD6244; ARRY-142886) or Placebo.
Groups:
- Placebo + Docetaxel 75 mg/m^2: Oral placebo BD and intravenous docetaxel on day 1 of every 21 day cycle
- Selumetinib 75 mg BD + Docetaxel 60 mg/m^2; Selumetinib 75 mg BD + Docetaxel 75 mg/m^2: Oral selumetinib BD and intravenous docetaxel on day 1 of every 21 day cycle
Period: Overall Study
Arm/Group | Placebo + Docetaxel 75 mg/m^2 | Selumetinib 75 mg BD + Docetaxel 60 mg/m^2 | Selumetinib 75 mg BD + Docetaxel 75 mg/m^2
Started | 43 | 85 | 84
Received Treatment | 43 | 84 | 84
Did Not Receive Treatment | 0 | 1 | 0
Completed | 0 | 0 | 0
Not Completed | 43 | 85 | 84
Not completed — Discontinued Selumetinib/Placebo | 37 | 77 | 75
Not completed — Ongoing Selumetinib/Pbo at data cut-off | 6 | 7 | 9
Not completed — Did not receive treatment | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Docetaxel 75 mg/m^2 | Selumetinib 75 mg BD + Docetaxel 60 mg/m^2 | Selumetinib 75 mg BD + Docetaxel 75 mg/m^2 | Total
Number analyzed (Participants) | 43 | 85 | 84 | 212
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (7.75) [47 to 76] | 62.4 (8.53) [41 to 84] | 60.4 (9.35) [38 to 79] | 61.8 (8.77) [38 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 26 | 61
  Male | 27 | 66 | 58 | 151
Race/Ethnicity, Customized [Number; unit: Participants]
  Black Or African American | 0 | 5 | 5 | 10
  Other | 2 | 0 | 1 | 3
  White | 41 | 80 | 78 | 199
KRAS Mutation Status at Baseline [Number; unit: Participants]
  KRAS no mutation detected (NMD) | 30 | 62 | 54 | 146
  KRAS mutation positive | 10 | 15 | 19 | 44
  KRAS mutation unknown | 3 | 8 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Median time from randomisation until the date of objective disease progression or death (by any cause in the absence of progression). Progression is defined using Response Evaluation Criteria in Solid Tumours (RECIST v1.1): >= 20% increase in the sum of diameters of Target Lesions (TL) and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of Non TLs or a new lesion.
Time Frame: Baseline and then every 6 weeks after randomization until objective disease progression, up to 29 months (at the time of the analysis)
Population: Full Analysis Set (All randomised patients). Progression events that do not occur within 14 weeks of the last evaluable assessement are censored and therefore excluded.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Placebo + Docetaxel 75 mg/m^2 | Selumetinib 75 mg BD + Docetaxel 60 mg/m^2 | Selumetinib 75 mg BD + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 36 | 75 | 69
Months | 4.3 [1.4 to 5.6] | 3.0 [1.4 to 5.4] | 4.2 [1.6 to 6.9]
Statistical Analysis 1: Comparison: Placebo + Docetaxel 75 mg/m^2 vs Selumetinib 75 mg BD + Docetaxel 60 mg/m^2; Test type: Non-Inferiority or Equivalence — A hazard ratio <1 favours selumetinib in combination with docetaxel; p = 0.584, Cox Proportional Hazards; Hazard Ratio (HR) = 1.12, 90% CI 2-sided [0.80 to 1.61]
Statistical Analysis 2: Comparison: Placebo + Docetaxel 75 mg/m^2 vs Selumetinib 75 mg BD + Docetaxel 75 mg/m^2; Test type: Non-Inferiority or Equivalence — A hazard ratio <1 favours selumetinib in combination with docetaxel; p = 0.690, Cox Proportional Hazards; Hazard Ratio (HR) = 0.92, 90% CI 2-sided [0.65 to 1.31]

2. Secondary Outcome: Overall Survival (OS)
Description: The time from randomisation until death due to any cause. Any subject not known to have died at the time of analysis will be censored based on the last recorded date on which the subject was known to be alive
Time Frame: Following progression, survival status was collected every 8 weeks until death, withdrawal of consent, or end of study, whichever occurred first, up to 29 months (at the time of the analysis)
Population: Full Analysis Set (All randomised patients)
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Placebo + Docetaxel 75 mg/m^2 | Selumetinib 75 mg BD + Docetaxel 60 mg/m^2 | Selumetinib 75 mg BD + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 43 | 85 | 84
Months | 11.5 [4.6 to 28.0] | 5.7 [3.1 to 12.4] | 7.7 [3.8 to 19.5]
Statistical Analysis 1: Comparison: Placebo + Docetaxel 75 mg/m^2 vs Selumetinib 75 mg BD + Docetaxel 60 mg/m^2; Test type: Non-Inferiority or Equivalence — A hazard ratio <1 favours selumetinib in combination with docetaxel; p = 0.126, Cox Proportional Hazards; Hazard Ratio (HR) = 1.43, 90% CI 2-sided [0.97 to 2.13]
Statistical Analysis 2: Comparison: Placebo + Docetaxel 75 mg/m^2 vs Selumetinib 75 mg BD + Docetaxel 75 mg/m^2; Test type: Non-Inferiority or Equivalence — A hazard ratio <1 favours selumetinib in combination with docetaxel; p = 0.485, Cox Proportional Hazards; Hazard Ratio (HR) = 1.18, 90% CI 2-sided [0.80 to 1.78]

ADVERSE EVENTS:
Arm/Group | Placebo + Docetaxel 75 mg/m^2 | Selumetinib 75 mg BD + Docetaxel 60 mg/m^2 | Selumetinib 75 mg BD + Docetaxel 75 mg/m^2
Serious Adverse Events (participants affected / at risk) | 16/43 | 40/84 | 38/84
Other Adverse Events (participants affected / at risk) | 38/43 | 80/84 | 83/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Docetaxel 75 mg/m^2 (N=43) | Selumetinib 75 mg BD + Docetaxel 60 mg/m^2 (N=84) | Selumetinib 75 mg BD + Docetaxel 75 mg/m^2 (N=84)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 4 (4)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1)
Performance status decreased (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 10 (13) | 4 (4)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 4 (4)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Docetaxel 75 mg/m^2 (N=43) | Selumetinib 75 mg BD + Docetaxel 60 mg/m^2 (N=84) | Selumetinib 75 mg BD + Docetaxel 75 mg/m^2 (N=84)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 20 (22) | 18 (21)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (4)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 3 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 10 (12) | 9 (26) | 17 (19)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (3)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3) | 3 (4)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Chorioretinal disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 3 (3)
Eye discharge (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 2 (5)
Eyelid pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 2 (2) | 2 (2) | 7 (7)
Noninfective conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1) | 3 (4)
Vision blurred (Eye disorders) | 0 (0) | 4 (4) | 3 (3)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 9 (12) | 6 (6)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5) | 3 (3) | 8 (9)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Breath odour (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Buccal mucosal roughening (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 16 (18) | 11 (13)
Dental cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 12 (21) | 41 (78) | 37 (65)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (10) | 6 (6) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (6)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip erosion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 10 (22) | 25 (33) | 23 (36)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral mucosal eruption (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Steatorrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 5 (7) | 11 (11) | 23 (33)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (13) | 20 (28) | 22 (27)
Asthenia (General disorders) | 2 (2) | 12 (12) | 13 (14)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 2 (2)
Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 4 (4) | 4 (4)
Fatigue (General disorders) | 13 (17) | 17 (21) | 26 (32)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 2 (2)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 3 (3)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 2 (2) | 3 (3)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1) | 7 (8)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 4 (4)
Oedema peripheral (General disorders) | 8 (10) | 16 (22) | 28 (38)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Performance status decreased (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (5) | 11 (15) | 11 (20)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Angular cheilitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2) | 6 (6)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 5 (5)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 4 (4) | 2 (2)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (5) | 1 (1)
Nosocomial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 3 (4) | 1 (1) | 1 (1)
Oral fungal infection (Infections and infestations) | 0 (0) | 4 (5) | 1 (2)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 1 (1) | 7 (9)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4) | 3 (3)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 5 (7)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (7) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (4) | 2 (2)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 3 (11) | 5 (11)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 2 (2)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 1 (2)
Ejection fraction decreased (Investigations) | 2 (2) | 4 (4) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 3 (3) | 6 (6)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Central obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10) | 21 (21) | 18 (20)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 4 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3) | 2 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (4) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (7) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6) | 9 (10)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (5) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4) | 2 (2)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 7 (7) | 5 (5) | 5 (5)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3) | 6 (6) | 8 (8)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 6 (6) | 3 (3)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (4) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 4 (4) | 4 (4)
Polyneuropathy (Nervous system disorders) | 1 (1) | 4 (4) | 3 (4)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (5) | 3 (3)
Sleep disorder (Psychiatric disorders) | 2 (3) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Costovertebral angle tenderness (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 5 (6)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal vein thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7) | 10 (10)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 12 (12) | 14 (15)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 4 (4)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (6) | 8 (9)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 7 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 5 (5)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 11 (11) | 15 (16)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (18) | 7 (9)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (10) | 16 (16)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 5 (6)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1)
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 9 (10) | 23 (26) | 29 (44)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (4) | 2 (2) | 10 (11)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 2 (2)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No